CLINICAL TRIAL: NCT05973825
Title: Immuno-virological Evaluation of Persons Living With HIV (PLWH) Who Initiated Anti-retroviral Treatment (ART) During Acute HIV Infection and of PLWH on Long Term ART
Brief Title: Immuno-virological Evaluation of Persons Living With HIV (PLWH)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Vrije Universiteit Brussel (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Centre Hospitalier Universitaire de Liege (Other); Universitair Ziekenhuis Brussel (Other); Université Libre de Bruxelles (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2023-0154
Record Dates: First submitted 2023-07-13; First posted 2023-08-03 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: HIV-1-infection; HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuno-virological evaluation of persons living with HIV (Experimental): Leucapheresis will be performed in HIV positive people making white blood cells available for in depth virological and immunological evaluation
  Interventions: Procedure: Leucapheresis

INTERVENTIONS:
Procedure: Leucapheresis — leucapheresis is a procedure in which a large amount of blood cells are obtained by an apheresis procedure

SUMMARY:
This is a dual arm (arm 1 and arm 2) multi-centric non-randomized (prospective) study.

Two new multicentric cohorts will be set up in 4 Belgian HIV reference centers (UZ Gent, UZ Brussel, University Hospital Liege and St. Pierre Hospital Brussels): cohort 1 will comprise PLWH in whom ART was initiated during acute HIV infection minimum 3 years ago but no more than 10 years ago (short-term ART cohort); cohort 2 will comprise PLWH on ART since >20 years (long-term ART cohort). Participants will be included based on suppressed viremia and uninterrupted ART since initiation. Participants will undergo one blood sampling and one leukapheresis. In and exclusion criteria are described below.

DETAILED DESCRIPTION:
This project aims to gain new knowledge and insights into the viral reservoir establishment and HIV Latency as well as to develop new powerful tools to study latency reversal, that will ultimately contribute to research into an HIV curative treatment.

The study objectives are

* To collect and store state of the art peripheral blood samples (60 vials of 50 X106 PBMC's) from two patient cohorts, 10 acute seroconverters and 10 long-term ART-treated patients .
* To characterize and compare the latent reservoir in blood samples from both cohorts as for the proviral genome, transcriptome, epigenome and T cell receptor level
* To perform an immunological profiling of infected cells.
* To evaluate available drugs that induce either a block-and-lock or a shock-and-kill in in vitro interventions using blood samples from both cohorts
* To accelerate the negative selection of transcriptionally competent proviruses in vitro and determine the role of the different determinants.
* To make all data available for the different partners and integrate all data acquired.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: short-term ART cohort

* Documented HIV-1 infection
* Able and willing to provide written informed consent
* Age = or >18 years and < 80 years
* ART started during a documented recent HIV-1 infection (acute HIV infection, defined as:

  * Clinical symptoms of acute seroconversion and incomplete Western Blot, or
  * Negative screening test within the past 6 months and incomplete Western Blot, or
  * Risk contact within the <3 months and presumable primo-infection with or without clinical symptoms and incomplete Western Blot.
* Being on ART since minimum 2 years and maximum 10 years
* Participants should have had a routine plasma viral load measurement at least once a year.
* Viral load < 40 or <50 copies/ml determined by the assay (used in the local centers) for at least 3 years (one blip < 200 copies/ml is allowed)
* Ability and willingness to have blood samples collected and stored for 20 years and used for various research purposes.
* Patients with HIV-1 subtype B are preferred for inclusion (as most of the complex assays are subtype B specific). However, if the investigators do not reach our target of 10 participants, patients infected with other subtypes will be allowed to enter the study. (Primers will subsequently be adapted to the patient-specific proviral sequences).

Cohort 2: long-term ART cohort

* Documented HIV-1 infection
* Able and willing to provide written informed consent
* Age = or >18 years and < 80 years
* Being on ART since at least 20 years
* ART should not have been started during a documented recent HIV-1 infection (acute HIV infection), defined as:

  * Clinical symptoms of acute seroconversion and incomplete Western Blot or
  * Negative screening test within the past 6 months and incomplete Western Blot or
  * Risk contact within <3 months and presumable primo-infection with or without clinical symptoms and incomplete Western Blot.
* Patients should have had a routine plasma viral load measurement at least once a year.
* Routine plasma viral load < 40 or <50 copies/ml determined by the assay used in the local centres for at least 20 years (one blip < 200 copies/ml is allowed if it occurred >10 years ago)
* Ability and willingness to have blood samples collected and stored for 20 years and used for various research purposes.
* Participants with HIV-1 subtype B are preferred for inclusion (as most of the complex assays are subtype B specific). However, if the investigators do not reach our target of 10 participants, patients infected with other subtypes will be allowed to enter the study. (Primers will subsequently be adapted to the patient-specific proviral sequences).

Exclusion Criteria:

* Previous or current history of opportunistic infection (AIDS defining events as defined in category C of the Centers for Disease Control and Prevention (CDC) clinical classification), consisting of chronic HIV-1 infection.
* Evidence of active Hepatitis B-virus (HBV) infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (= HBV antigen or viral load negative and positive HBV surface antibody).
* Evidence of active HCV infection (HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry).
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease.
* Current cancer.
* History of HIV-related thrombocytopenia.
* Pregnancy or breastfeeding.
* Any condition, including preexisting psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant.
* Abnormal results of standard of care laboratory tests:

  1. Confirmed haemoglobin <11g/dl for women and <12 g/dl for men
  2. Confirmed platelet count <100 000/µl *
  3. Confirmed neutrophil count <1000/μl
  4. Confirmed Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>10x upper limit of normal (ULN)
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-07-12 (Estimated); Study Completion 2029-07-12 (Estimated)

PRIMARY OUTCOMES:
Information on virological aspects of people on long term ART versus people treated during recent infection | 3 years
  Intact proviral deoxyribonucleic acid (DNA) assay quantified by digital Polymerase Chain Reaction (pcr)

CONTACTS AND LOCATIONS:
Overall Officials: Linos vandekerckhove, Principal Investigator — UZ Gent
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium